CLINICAL TRIAL: NCT00261703
Title: Randomized Phase III Trial Comparing Induction Chemotherapy With Cisplatin/5-fluorouracil (PF) or Docetaxel/Cisplatin/5-fluorouracil (TPF) Plus Chemoradiotherapy (CRT) Versus CRT Alone as First-line Treatment or Unresectable Locally Advanced Head and Neck Cancer (LAHNC).
Brief Title: Docetaxel in Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976F_2503
Record Dates: First submitted 2005-12-02; First posted 2005-12-05 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Head and Neck Neoplasms
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy

ARMS (3):
- 1 (Experimental): (Docetaxel + Cisplatin + 5-FU) + Cisplatin + Radiotherapy
  Interventions: Drug: Docetaxel, Cisplatin, 5-fluorouracil (5-FU), radiotherapy
- 2 (Experimental): (Cisplatin + 5-FU) + Cisplatin + Radiotherapy
  Interventions: Drug: Cisplatin, 5-fluorouracil (5-FU), radiotherapy
- 3 (Experimental): Cisplatin + Radiotherapy
  Interventions: Other: Cisplatin + radiotherapy

INTERVENTIONS:
Drug: Docetaxel, Cisplatin, 5-fluorouracil (5-FU), radiotherapy — Docetaxel 75 mg/m2, Day 1 of the cycle + Cisplatin 75 mg/m2 Day 1 + 5-FU 750 mg/m2/day in 24-h continuous infusion for 5 days. 3 cycles will be administered, every 21 days, before the local-regional treatment (same as control group)
  Arms: 1
Drug: Cisplatin, 5-fluorouracil (5-FU), radiotherapy — Cisplatin 100 mg/m2 Day 1, 5-FU 1000 mg/m2/day in 24-h continuous infusion for 5 consecutive days. 3 cycles will be administered every 21 days, before the local-regional treatment (same as control group)
  Arms: 2
Other: Cisplatin + radiotherapy — Cisplatin 100 mg/m2 on days 1, 22 and 43 simultaneously with radiotherapy (2 Gy x 1/day, 5 days per week for 7 weeks-tumor- and 2 Gy x 1/day, 5 days per week for 6 weeks- lymph nodes)
  Arms: 3

SUMMARY:
Primary Objective:

* Phase II: To determine the best treatment scheme (TPF vs. PF).
* Phase III: To compare the time to progression and the treatment failure at the 3 arms.

Secondary objectives:

* To evaluate the safety at the 3 arms.
* To compare the progression , overall survival and locoregional control at the 3 arms.

ELIGIBILITY:
Inclusion Criteria:

* Head and Neck cancer locally advanced (oral cavity, oropharynx, hypopharynx or larynx) but without evident metastasis.
* Inoperable tumor after revision by a multidisciplinary oncology team.
* Proved epidermoid carcinoma.
* ECOG = 0-1
* Good hematologic function (i.e, hemoglobin > 10 g/dl, ...)
* Good hepatologic function
* Good renal function

Exclusion Criteria:

* Pregnant or breast-feeding women. Potential child-bearing women should use an effective conceptive method and should have a negative pregnancy test at least the week before entering the study.
* Nasopharynx, nasal cavity and paranasal sinusitis will be excluded
* Previous chemotherapeutic or radiotherapeutic treatment for this disease.
* Previous or current neoplasms in other locations, except in situ cervicouterine cancer properly treated or basal cell or squamous cell carcinoma
* Symptomatic peripheral neuropathy
* Other clinical severe diseases
* Concomitant treatment with corticoids within 6 months prior to inclusion.
* Concomitant treatment with any other neoplastic therapy
* Previous treatment for current disease.
* Loss of weight greater than 10% within the last 3 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2002-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Phase II: Clinical objective response rate, at the end of inducted chemotherapy (groups A and B) and at the end of combined treatment (groups A, B and C). | 16 weeks
Phase III: Surveillance with no progression after two years. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: JOSÉ Mª TABOADA, Study Director — Sanofi
Locations (2):
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Barcelona, Spain

REFERENCES:
- [Derived] Hitt R, Iglesias L, Lopez-Pousa A, Berrocal-Jaime A, Grau JJ, Garcia-Giron C, Martinez-Trufero J, Guix M, Lambea-Sorrosal J, Del Barco-Morillo E, Leon-Vintro X, Cunquero-Tomas AJ, Baste N, Ocana A, Cruz-Hernandez JJ; the Spanish Head and Neck Cancer Cooperative Group (TTCC). Long-term outcomes of induction chemotherapy followed by chemoradiotherapy vs chemoradiotherapy alone as treatment of unresectable head and neck cancer: follow-up of the Spanish Head and Neck Cancer Group (TTCC) 2503 Trial. Clin Transl Oncol. 2021 Apr;23(4):764-772. doi: 10.1007/s12094-020-02467-8. Epub 2020 Aug 14. PMID 32797376
- [Derived] Hitt R, Grau JJ, Lopez-Pousa A, Berrocal A, Garcia-Giron C, Irigoyen A, Sastre J, Martinez-Trufero J, Brandariz Castelo JA, Verger E, Cruz-Hernandez JJ; Spanish Head and Neck Cancer Cooperative Group (TTCC). A randomized phase III trial comparing induction chemotherapy followed by chemoradiotherapy versus chemoradiotherapy alone as treatment of unresectable head and neck cancer. Ann Oncol. 2014 Jan;25(1):216-25. doi: 10.1093/annonc/mdt461. Epub 2013 Nov 19. PMID 24256848